CLINICAL TRIAL: NCT03501849
Title: Improving Complete Resection Rates of 4-20mm Adenomas Using Cold Snare Polypectomy
Brief Title: Cold Snare Polypectomy
Acronym: Cold-Snare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17.296
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2018-04

CONDITIONS: Colorectal Cancer; Colon Adenoma
Keywords: Cancer prevention; Cancer detection; Colonoscopy; Polypectomy; Cold Snare
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polypectomy using a cold snare (Experimental): Polypectomy by cold-snare technique
  Interventions: Device: Polypectomy using a cold snare

INTERVENTIONS:
Device: Polypectomy using a cold snare — Polypectomy by cold-snare technique

SUMMARY:
During colonoscopy, the endoscopist will document prospectively all polyps detected and note the size, location and morphology. Polyps of 4-20 mm will be removed only in accordance with the method the cold snare. Afterwards, the remaining tissues could be observed with an imaging technology called Optivista with an injection of 10-50 ml of saline solution (if required) to improve visibility of the tissues. The endoscopist will continue to remove the remaining polyp tissue (with a snare or forceps) until there are no more visible polyp tissues. Biopsies from the polyp resection site will be sent to the laboratory for analysis to confirm the complete resection.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a major global disease affecting more than 1 million people worldwide and the majority of colon cancers develop from adenomas. The purpose of endoscopic cancer prevention is the detection and removal of these precancerous adenomatous polyps. However, polyps between 4-20 mm are incompletely eliminated in about 10% of cases, which is one of the main risk factors for patients to develop post-colonoscopy cancers. The polypectomy with cold snare showed promising results for complete adenoma resection rates for polyps up to 9 mm.

The hypotheses is that polypectomy with cold snare could be a standard approach for polyps up to 20 mm and could improve the rates of complete resection of the adenoma.

All eligible patients to undergo colonoscopy will be considered for the project.

Patients will be identified from the colonoscopy appointment lists at the CHUM. During colonoscopy, the endoscopist will document prospectively all polyps detected and note the size, location and morphology. All polyps will be removed during the procedure and will be sent to the laboratory as recommended in current clinical practice. Polyps of 4-20 mm will be removed only in accordance with the method the cold snare. Afterwards, the remaining tissues could be observed with an imaging technology called Optivista with an injection of 10-50 ml of saline solution (ir required) to improve visibility of the tissues. Optivista is an imaging technique based that uses a light filter for endoscopic optical diagnosis where light of specific blue and green wavelengths is used to enhance the surface and vascular patterns of the polyp surface mucosa. The intestinal mucosa will be carefully examined and the endoscopist will continue to remove the remaining polyp tissue (with a snare or forceps) until there are no more visible polyp tissues. Biopsies from the polyp resection site will be sent to the laboratory for analysis to confirm the complete resection.

Telephone follow-up will be done 14 days after the procedure to report possible side effects occurred.

The rate of incomplete resection of all adenomatous polyps resected in the cold snare will be determinate after completion of this project. The confidence interval will first be calculated using the exact confidence limits of Clopper-Pearson, considering all adenomatous polyps. An additional analysis will also be performed with a model of estimation equations (GEE) based on the binomial distribution to obtain standard errors taking into account the correlation with the patient.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 45 to 80 years
* Indication for full colonoscopy

Exclusion Criteria:

* Known inflammatory bowel disease
* Active colitis
* Coagulopathy
* Familial polyposis syndrome
* Poor general health defined as an ASA class > 3
* Emergency colonoscopies defined as patients with evidence of hemodynamic instability and/or ongoing active GI bleeding and/or intensive care requirements.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Incomplete resection rate (in percentage) | 2 years
  Incomplete resection rate as defined by any adenomatous polyp tissue found in at least one marginal biopsies

SECONDARY OUTCOMES:
Number of immediate bleeding complication (numerical) | 2 years
  Defined as bleeding requiring endoscopic intervention either during colonoscopy/ polypectomy, or requiring an immediate second intervention such as surgery and/or hospital admission
Number of delayed bleeding complications (numerical) | 2 years
  Defined as bleeding after the end of the initial procedure until 30 days later, requiring a second endoscopic intervention or another intervention such as surgery and/or hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Daniel von Renteln, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Montréal (CHUM)
Locations (1):
- Centre Hospitalier Universitaire de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] von Renteln D, Djinbachian R, Benard F, Barkun AN, Bouin M, Bouchard S, Deslandres E, Panzini B, Sidani S, Leduc R, Jobse BC, Pohl H. Incomplete resection of colorectal polyps of 4-20 mm in size when using a cold snare, and its associated factors. Endoscopy. 2023 Oct;55(10):929-937. doi: 10.1055/a-1978-3277. Epub 2022 Nov 14. PMID 36377124